CLINICAL TRIAL: NCT06942871
Title: Non-Invasive Lung Water Monitoring Guided by Remote Dielectric Sensing Technology in the Management of Patients With Pulmonary Hypertension
Brief Title: Non-Invasive Lung Water Monitoring in Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ReDS in PAH
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung fluid: The measurement of ReDS values was performed with the patient in a seated position and under normal breathing conditions. It was conducted on the morning of the second day following admission or at the end of an outpatient visit. The device's sensors or vest were properly placed on the patient's chest to ensure good contact between the sensors and the skin. Upon initiating the measurement program, the device emitted low-power electromagnetic signals that passed through the thorax and lungs. It measured the dielectric constant (impedance) of the lungs and calculated the percentage of lung fluid. The manufacturer-recommended normal range is between 20% and 35%. The entire measurement process took approximately 45 seconds.
  Interventions: Device: Remote Dielectric Sensing

INTERVENTIONS:
Device: Remote Dielectric Sensing — The lung fluid monitor Remote Dielectric Sensing (ReDS™) is the world's first non-invasive device for heart failure monitoring and management. It directly reflects lung fluid content by measuring changes in thoracic dielectric constants, with a detection range of 15% ~ 60%. The device can sensitively identify pathological states ranging from mild compensation to severe pulmonary edema. ReDS™ technology cannot directly measure pulmonary artery pressure, but changes in lung fluid content may indirectly reflect disease progression in certain types of pulmonary hypertension.

SUMMARY:
The investigators conducted a prospective, convenience-sampled observational pilot study, enrolling adult patients with pulmonary hypertension who were either outpatients or inpatients in the cardiology department of our hospital. The measurement of Remote Dielectric Sensing (ReDS) values was performed by ReDS™ Pro. Data were collected using the electronic medical record system of our hospital. Participants were followed up within 6 months after discharge. The primary endpoints included all-cause mortality or clinical deterioration related to pulmonary hypertension.

DETAILED DESCRIPTION:
The investigators conducted a prospective, convenience-sampled observational pilot study, enrolling adult patients with pulmonary hypertension who were either outpatients or inpatients in the cardiology department of our hospital. The measurement of Remote Dielectric Sensing (ReDS) values was performed by ReDS™ Pro. Data were collected using the electronic medical record system of our hospital. Participants were followed up within 6 months after discharge. The primary endpoints included all-cause mortality or clinical deterioration related to pulmonary hypertension. Data were collected using the electronic medical record system of our hospital, including demographics, clinical diagnoses, past medical history, ancillary examinations and laboratory test, surgical procedures, and medication use. Treatment and management of participants were in accordance with guideline recommendations. Participants were followed up by telephone or outpatient visits within 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤85 years, with no gender restriction;
* Hemodynamic confirmation of PH via right heart catheterization (RHC) (mean pulmonary arterial pressure [mPAP] > 20 mmHg).

Exclusion Criteria:

* Thoracic deformities or injuries precluding proper device fit (e.g., severe scoliosis, flail chest);
* Inability to use the ReDS™ Pro non-invasive lung fluid monitor due to physical characteristics (height <155 cm or >190 cm; body mass index [BMI] <22 kg/m² or >39 kg/m²);
* Prior implantation of a left ventricular assist device or cardiac transplantation;
* Congenital cardiac anomalies or intrathoracic masses affecting right lung anatomy;
* Hemodynamic profiles inconsistent with PH.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients with PH who were admitted to the Department of Cardiology at Zhongshan Hospital, Fudan University, between April 2024 and March 2025 were prospectively enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
all-cause mortality or clinical deterioration related to PH | The follow-up period is up to March 31, 2025.
  1) all-cause death or lung transplantation; 2) rehospitalization due to PH-related heart failure; 3) worsening of WHO cardiac functional class.

CONTACTS AND LOCATIONS:
Overall Officials: Dandan CHEN, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humbert M, Kovacs G, Hoeper MM, Badagliacca R, Berger RMF, Brida M, Carlsen J, Coats AJS, Escribano-Subias P, Ferrari P, Ferreira DS, Ghofrani HA, Giannakoulas G, Kiely DG, Mayer E, Meszaros G, Nagavci B, Olsson KM, Pepke-Zaba J, Quint JK, Radegran G, Simonneau G, Sitbon O, Tonia T, Toshner M, Vachiery JL, Vonk Noordegraaf A, Delcroix M, Rosenkranz S; ESC/ERS Scientific Document Group. 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Heart J. 2022 Oct 11;43(38):3618-3731. doi: 10.1093/eurheartj/ehac237. No abstract available. PMID 36017548
- [Background] Bensimhon D, Alali SA, Curran L, Gelbart E, Garman DWV, Taylor R, Chase P, Peacock WF. The use of the reds noninvasive lung fluid monitoring system to assess readiness for discharge in patients hospitalized with acute heart failure: A pilot study. Heart Lung. 2021 Jan-Feb;50(1):59-64. doi: 10.1016/j.hrtlng.2020.07.003. Epub 2020 Jul 20. PMID 32703623
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e876-e894. doi: 10.1161/CIR.0000000000001062. Epub 2022 Apr 1. PMID 35363500
- [Derived] Chen D, Tian D, Jin Q, Zhang L, Zhang X, Li M, Pan W, Lv Q, Zhou D, Ge J, Guan L. The potential of non-invasive remote dielectric sensing in predicting short-term prognosis of patients with pulmonary hypertension. BMC Pulm Med. 2025 Oct 8;25(1):460. doi: 10.1186/s12890-025-03922-4. PMID 41063151